CLINICAL TRIAL: NCT01808066
Title: GroundsKeeper: A Qualitative Study of Applied Game-based Interactives in Special Education Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CogCubed, Corp (Industry)
Collaborators: Ohio University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12X226; 12X226 (Other: Ohio University IRB)
Record Dates: First submitted 2013-03-06; First posted 2013-03-11 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder; Pervasive Developmental Disorder; Asperger's Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Child Development Disorders, Pervasive; Asperger Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Play Groundskeeper (Experimental): This study will employ design-based research models (Laurel, 2003) to the executive-functioning training game GroundsKeeper by CogCubed; we will assess the quality of digital designs for learning (Barab & Squire, 2004) using established qualitative data collection to analyze game play and player reaction over a three week period of time. We will assess the participants for their ability to stay engaged in play by observing their engagement in the game, time played, frequency of play, and the ability to complete a session over the course of three weeks while in school.
  Interventions: Device: Groundskeeper

INTERVENTIONS:
Device: Groundskeeper — Groundskeeper is a product developed for helping players develop skills to increase focus and attention. The game is played on small Sifteo Cubes that have sensors that react to you and each other. There are new games that might help children with ADHD and Autism learn to better focus and keep attention on a task.
  Other Names: Executive Function Training Game

SUMMARY:
The purpose of this study is to examine the use of, and reaction to, one particular software application(GroundsKeeper) delivered on unique platform - Sifteo cubes (www.sifteo.com). The hypothesis is that the use of these devices will increase engagement, motivation, interest, and have perceived benefits to users with unique attention-limiting cognitive disabilities. How does the observation of and user feedback from gameplay reveal areas of improvement for the game, strengths, and perceptions of value among the players and adults?

DETAILED DESCRIPTION:
Primarily the investigators seek to observe and interview participants over a three-week period of time to assess their ongoing interest and the perceived effects of regular play segments each day (10-20 minutes each). Data will be collected in pre/post interviews, teacher journals, and observation of pre/post play sessions.

These new hands-on digitized cubes are motion sensitive blocks that are capable of interactively reacting to each other and motion applied to them. The game GroundKeeper makes use of these cubes to use auditory and visual stimuli to provide distractors during play apart from the goal of the game. The investigators expect that play will encourage attention in players and are interested to see what players and their teachers/parents perceive the effects to be.

The investigator's goal is not to measure actual attention rates and times of the students, but the subjective observations of players' engagement with the devices, motivation to play the game, interest initially and over time, and perceived effect of the game on attention. This type study is commonly known as 'play-testing' a software product with the target audience; a process refined as "design-based research" in academia (Laurel, 2003) and used for assessing the quality of digital designs for learning (Barab & Squire, 2004) and using data to improve them. This study will be a qualitative counter-balance to the quantitative work being done separately by the University of Minnesota (Under Dr. Srivastava), using clinical and computer based diagnostics and data mining respectively on the same product.

Digital tools are facilitating both traditional and '21st century skills' via new information and communication technologies for knowledge work, thinking, learning, and leading digital lifestyles (p. 23) (Trilling & Fadel, 2009). Further there is growing evidence these skills, along with traditional literacies are being learned by using digital applications (Gee, 2007; Squire & Barab, 2004; Steinkuehler & Duncan, 2008). Early evidence that digital tools can 'amplify' learning activity shows potential for digital technology to beneficial even if 'played' or used 'in the wild' (Squire & Dikkers, 2012). This study seeks to further explore learning attributes of a digitally mediated learning experience designed for a particular learning goal.

Additionally, current diagnostic aids, used in treating attention capacity for Attention Deficit Hyperactivity Disorder (ADHD) and Autism, are currently expensive, time intensive, and provide little information about accessory movements in response to a stimulus. One in ten children, ages 5 to 17, has been diagnosed with ADHD; and the number of kids with autism has increased 78% in the last ten years http://www.cnn.com/2012/03/29/ health/autism/index.html). This study will seek to assess the accessibility and usability of software that seeks to help shape attention strategies through play and 'fun' learning for both ADHD and Autistic children that struggle with attention. If effective this could be a valuable and affordable option for educational institutions to serve these learners.

This study seeks to aid CogCubed in improved design for their game that will improve its' ability to engage, motivate, and retain player interest over time.

ELIGIBILITY:
Inclusion Criteria:

* Attention Deficit Hyperactivity Disorder
* Autism Spectrum Disorder
* Pervasive Developmental Disorder
* Asperger's Disorder
* Cognitive Disabilities

Exclusion Criteria:

* Subject does not have cognitive disabilities, Attention Deficit Hyperactivity Disorder or Autism Spectrum Disorders

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seann Dikkers, PhD, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

REFERENCES:
- [Background] Trilling, Bernie, & Fadel, Charles. (2009). 21 Century Skills: Learning for Life in our Times. San Francisco, CA: Jossey-Bass.
- [Background] Steinkuehler, C., & Duncan, S. (2008). Scientific Habits of Mind in Virtual Worlds. Journal of Science Education and Technology, 17(6), 530-543. doi: Doi 10.1007/S10956-008-9120-8
- [Background] Squire, K., & Dikkers, S. (2012). Amplifications of learning: Use of mobile media devices among youth. Convergence: The International Journal of Research into New Media Technologies, OnlineFirst. http://con.sagepub.com/content/early/2012/02/15/1354856511429646 doi:10.1177/1354856511429646.
- [Background] Squire, K., & Barab, S. (2004). Replaying history: Engaging urban undeserved students in learning world history. Paper presented at the 6th international conference on Learning sciences, Los Angeles, CA.
- [Background] Gee, J. P. (2007). What Video Games have to Teach us about Learning and Literacy. New York, NY: Palgrave Macmillan
- [Background] Barab, S. and K. Squire (2004).
- [Background] Laurel, B., Ed. (2003). Design Research: Methods and Perspectives. Cambridge, MA, The MIT Press.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: 21 participants with ADHD who underwent the intervention for 3 weeks, played for 20 minutes at a time at school.
Period: Overall Study
Arm/Group | Treatment Group
Started | 21
Completed | 6
Not Completed | 15
Not completed — Withdrawal by Subject | 15

BASELINE CHARACTERISTICS:
Population: students at school grades K-6
Groups:
- Play Groundskeeper: This study will employ design-based research models (Laurel, 2003) to the executive-functioning training game GroundsKeeper by CogCubed; we will assess the quality of digital designs for learning (Barab & Squire, 2004) using established qualitative data collection to analyze game play and player reaction over a three week period of time.
  Groundskeeper: Groundskeeper is a product developed for helping players develop skills to increase focus and attention. The game is played on small Sifteo Cubes that have sensors that react to you and each other. There are new games that might help children with ADHD and Autism learn to better focus and keep attention on a task.
Arm/Group | Play Groundskeeper
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 8 [5 to 11]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Increase/Improvement in Focusing
Description: Researchers will observe and record data during the first play session. Over the three weeks, teachers/support staff will be asked to observe players each day and record their observations as needed in a journal. These observations will measure their improvement in their ability to focus by assessing their engagement, time played, frequency of play, ability to complete a session and ability to start and finish a session. At the end of three weeks, researchers will attend the final play session and record observations in writing.
Time Frame: 3 weeks
Measure: Number; unit: participants
Arm/Group | Play Groundskeeper
Number analyzed (Participants) | 21
participants | 6

2. Secondary Outcome: Number of Participants Identified as Attentive, Interested and Motivated Via Pre Interview
Description: Researchers will conduct interviews with players and collect all notes/journals recorded. Specific questions will be asked about their perception of their attention, interest and motivation to play the game. Example of questions included if they enjoyed playing the game, if they wanted to play the game and if they have trouble focusing during the game. Was it too long? Themes of the answers will be identified by researchers as a qualitative measure of interest.
Time Frame: Day 1
Population: participants in a school who underwent the intervention for 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
Participants | 21

3. Other Pre Specified Outcome: Number of Participants by Teachers Identified as Attentive, Interested and Motivated Via Pre Interview
Description: Researchers will conduct interviews with teachers and collect all notes/journals recorded. Specific questions will be asked about their perception of their attention, interest and motivation to play the game. Example of questions included if they enjoyed playing the game, if they wanted to play the game and if they have trouble focusing during the game. Was it too long? Themes of the answers will be identified by researchers as a qualitative measure of interest.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
Participants | 21

4. Other Pre Specified Outcome: Number of Participants Identified as Interested and Improved Quality of Life in Classroom Via Post Test Interview
Description: After playing game for three weeks, researchers will interview participants about their interest in the game and changes in quality of life (no forms).
Time Frame: Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Play Groundskeeper
Number analyzed (Participants) | 21
Participants | 21

5. Other Pre Specified Outcome: Number of Participants Identified by Teachers as Attentive, Interested and Motivated Following Testing Via Post Test Interview
Description: Researchers will ask teachers for qualitative feedback once participants have completed game play about interest in using the game and any improvements to be made. Did they think the game was interactive. Would they use the game again? Do they think the students were able to maintain their interest?
  Number of Participants identified as attentive, interested and motivated via pre interview
Time Frame: Day 21
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
Participants | 21

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
Technical difficulties resulting from firewall at school affected set up time, difficulty with log in instructions and the cubes sliding on desktops.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No